CLINICAL TRIAL: NCT01583465
Title: Open Label, Randomized, Blinded Study to Evaluate the Efficacy of Aquamantys System for Reducing the Transfusion Requirements Associated With the Anterior-Supine Intermuscular (ASI) Approach for Total Hip Arthroplasty (THA)
Brief Title: Efficacy of Aquamantys for Reducing Transfusions With Anterior Supine Intermuscular Approach Total Hip Arthroplasty
Acronym: Aquamantys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Implant Surgeons, Inc. (Other)
Collaborators: Medtronic (Industry); Mount Carmel Health System (Other)
Responsible Party: Principal Investigator, Keith R. Berend, Principal Investigator, Joint Implant Surgeons, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20091312
Record Dates: First submitted 2012-04-18; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis, Hip; Joint Deformities, Acquired; Hip Dislocation, Congenital; Osteonecrosis; Arthritis, Rheumatoid
Keywords: randomized controlled trial; Blood loss, surgical; Blood loss, postoperative; Wound healing
MeSH Terms: conditions — Osteoarthritis, Hip; Joint Deformities, Acquired; Hip Dislocation, Congenital; Osteonecrosis; Arthritis, Rheumatoid; Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Ultraviolet Therapy; Electrocoagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aquamantys Malleable Bipolar Sealer (Experimental): In 100 patients randomly assigned, primary total hip arthroplasty via an anterior supine intermuscular approach will be performed with the assistance of the Aquamantys Malleable Bipolar Sealer with Light.
  Interventions: Device: Aquamantys
- Standard Treatment (Active Comparator): 100 patients randomly assigned will undergo primary total hip arthroplasty via the anterior supine intermuscular approach performed with the assistance of standard electrocautery.
  Interventions: Device: standard electrocautery (Bovie)

INTERVENTIONS:
Device: Aquamantys — Primary THA via the ASI approach will be performed using the Aquamantys Malleable Bipolar Sealer. The Aquamantys is a bipolar device that combines radio-frequency energy and saline to gently reach targeted tissue and provide a biomechanical seal. The saline acts as a conduit to allow the energy to penetrate the tissue from 1 to 2 mm where the collagen is transformed thus providing the seal. The saline also helps cool the tissue which allows for gentle handling of tissue, eliminating the black char that is a port for infection. The surgeon uses the Aquamantys to assist in tissue dissection, cauterize vessels, and to pre-treat fat pad in front of capsule prior to excision, to treat the entire anterior hip capsule prior to excision, treat oozing bone surfaces not covered by an implant.
  Other Names: Aquamantys Malleable Bipolar Sealer with Light; 21 CFR 878.4400; Electrosurgery Bipolar Sealer
  Arms: Aquamantys Malleable Bipolar Sealer
Device: standard electrocautery (Bovie) — Primary total hip arthroplasty via an anterior supine intermuscular approach will be performed with the assistance of standard electrocautery. The electrocautery is used in tissue dissection and to cauterize bleeding vessels.
  Other Names: electrocautery; Bovie
  Arms: Standard Treatment

SUMMARY:
The purpose of this study is to establish whether or not there is a clinical advantage to the use of Aquamantys® System from Medtronic Advanced Energy (formerly Salient Surgical Technologies) in patients undergoing primary total hip arthroplasty via the anterior supine intermuscular surgical approach in terms of blood loss, transfusion and wound healing. Wound healing will be assessed by a blinded observer and based upon a simple and subjective criteria: a) as expected, b) better than expected or c) worse than expected. The blinded observer is experienced in the care of the surgical patient and wound evaluation.

DETAILED DESCRIPTION:
To establish in a randomized, blinded study whether or not there is a clinical advantage to the use of Aquamantys® System from Medtronic Advanced Energy (formerly Salient Surgical Technologies) in patients undergoing primary total hip arthroplasty via the anterior supine intermuscular surgical approach in terms of blood loss, transfusion and wound healing based on early collected data. Data will be analyzed using StatsDirect in standard fashion to elucidate any difference between control and treatment groups. Wound healing will be assessed by a blinded observer and based upon a simple and subjective criteria: a) as expected, b) better than expected or c) worse than expected. The blinded observer is experienced in the care of the surgical patient and wound evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary unilateral total hip arthroplasty via the anterior supine intermuscular approach
* Patient is willing and able to complete all follow-up visits at 6 weeks and 1 year

Exclusion Criteria:

* Patients with pre-existing known coagulopathy
* Patients on chronic Coumadin (Warfarin) therapy
* Patients receiving erythropoietin therapy for anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Perioperative Change in Hemoglobin Level | From up to 30 days preoperative through postoperative day 1
  All patients will undergo routine lab work perioperatively. No additional studies will be necessary for this protocol. Hemoglobin level will be first measured preoperatively at the time of preadmission testing, which must be performed not more than 30 days prior to surgery, and then measured on postoperative day one. The two levels will be compared to assess the decrease in hemoglobin level resulting from the surgical intervention.
Perioperative Blood Transfusion Requirement | From the beginning of surgical intervention to hospital discharge, which averages 2 days and may be up to 1 week postoperative
  Perioperative blood transfusion requirements will be recorded, including transfusions administered during the surgical intervention and throughout the acute hospital stay.
Perioperative Blood Loss | From beginning of surgical intervention through hospital discharge, which averages 2 days and may be up to 1 week
  Anesthesia and nursing records will be monitored for blood loss intraoperatively, and postoperatively via drain output. Drains will be pulled daily at 0600 and measured.

SECONDARY OUTCOMES:
The development of complications in the wound, either as an inpatient or after discharge | Wound evaluations will occur each postoperative day in hospital (average 2 days and up to 1 week), at 6 weeks, and 1 year.
  Wound care will be evaluated by a designee who will be blinded to the randomization. Wound will be evaluated for drainage, erythema, and ecchymosis. Additionally, the wound healing will be scored as: Healing better than expected, As expected, or Worse than expected. Wound evaluations will occur each postoperative day in hospital (average 2 days), at 6 weeks, and 1 year.
Length of stay | From admission through hospital discharge (average 2 days, up to 1 week)
  Length of acute hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Berend, MD, Principal Investigator — Joint Implant Surgeons, Inc.
Locations (1):
- Joint Implant Surgeons, Inc., New Albany, Ohio, United States

REFERENCES:
- [Result] Barsoum WK, Klika AK, Murray TG, Higuera C, Lee HH, Krebs VE. Prospective randomized evaluation of the need for blood transfusion during primary total hip arthroplasty with use of a bipolar sealer. J Bone Joint Surg Am. 2011 Mar 16;93(6):513-8. doi: 10.2106/JBJS.J.00036. PMID 21411700
- [Result] Zeh A, Messer J, Davis J, Vasarhelyi A, Wohlrab D. The Aquamantys system--an alternative to reduce blood loss in primary total hip arthroplasty? J Arthroplasty. 2010 Oct;25(7):1072-7. doi: 10.1016/j.arth.2009.10.008. Epub 2010 Jan 22. PMID 20097039
- [Result] Mankin KP, Moore CA, Miller LE, Block JE. Hemostasis with a bipolar sealer during surgical correction of adolescent idiopathic scoliosis. J Spinal Disord Tech. 2012 Jul;25(5):259-63. doi: 10.1097/BSD.0b013e3182334ec5. PMID 21964452
- [Result] Morris MJ, Berend KR, Lombardi AV Jr. Hemostasis in anterior supine intermuscular total hip arthroplasty: pilot study comparing standard electrocautery and a bipolar sealer. Surg Technol Int. 2010 Oct;20:352-6. PMID 21082586
- [Result] Marulanda GA, Ulrich SD, Seyler TM, Delanois RE, Mont MA. Reductions in blood loss with a bipolar sealer in total hip arthroplasty. Expert Rev Med Devices. 2008 Mar;5(2):125-31. doi: 10.1586/17434440.5.2.125. PMID 18331175
- [Result] Marulanda GA, Ragland PS, Seyler TM, Mont MA. Reductions in blood loss with use of a bipolar sealer for hemostasis in primary total knee arthroplasty. Surg Technol Int. 2005;14:281-6. PMID 16525984
- [Result] Marulanda GA, Krebs VE, Bierbaum BE, Goldberg VM, Ries M, Ulrich SD, Seyler TM, Mont MA. Hemostasis using a bipolar sealer in primary unilateral total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2009 Dec;38(12):E179-83. PMID 20145794
- See also: Manufacturer's website; Related Info — http://www.salientsurgical.com/
- See also: Related info; animated sequence — http://www.youtube.com/watch?v=s5O91NjEuCM
- See also: Related info — http://www.whichmedicaldevice.com/by-manufacturer/49/293/aquamantys-system